CLINICAL TRIAL: NCT05972733
Title: Phase 2, Single-arm, Open-label Trial for Serologic Assay Validation, Proficiency Testing, Safety and Immunogenicity of the Intramuscular HIL-214 Norovirus Vaccine in Adults Aged 18 to 49 Years
Brief Title: Serologic Assay Validation and Proficiency Testing of HIL-214 in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HilleVax (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NOR-215
Record Dates: First submitted 2023-07-11; First posted 2023-08-02 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Intervention Model Description: Single-arm, Open-label Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Arm Study (Experimental): One dose given to all participants
  Interventions: Biological: HIL-214

INTERVENTIONS:
Biological: HIL-214 — HIL-214

SUMMARY:
The purpose of this trial is to obtain serum for proficiency testing to confirm assay validity is maintained following the dosing of adults with a pediatric dose of HIL-214.

DETAILED DESCRIPTION:
This single-arm trial serves to obtain serum for proficiency testing to confirm assay validity is maintained. Exploratory aspects of this trial include evaluating additional assays used for the assessment of immune responses to HIL-214 in peripheral-blood samples. Given the large volume of blood required, the pediatric dose will be tested in healthy adults. The main scientific rationale for the trial is to identify immune assays that can assess the generation of serum antibodies or cell-mediated immunity (CMI) specific to norovirus strains not represented in the HIL-214 vaccine (i.e. cross-reactivity).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 49 years, inclusive.
* Individuals who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
* The individual signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to regulatory requirements.
* Individuals willing and able to comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

* Females who are pregnant or breastfeeding.
* Gastroenteritis within 14 days before planned dosing (can warrant delay of trial vaccine administration).
* Known hypersensitivity or allergy to any of the HIL-214 components (including excipients).
* Known or suspected impairment/alteration of immune function, including history of any autoimmune disease or neuro-inflammatory disease.
* Any serious chronic or progressive disease (including hepatitis B or C).
* Previous exposure to an experimental norovirus vaccine.
* Subject or subject's first-degree relatives are involved in the trial conduct.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pennisula Research Associates, Rolling Hills Estates, California
  - Clinical Research Atlanta, Stockbridge, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the trial at 2 investigative sites in the United States from 01 August 2023 to 10 November 2023.
Pre-assignment Details: Healthy volunteers were enrolled in 1 treatment arm and received a single dose of HIL-214, a norovirus vaccine comprising 50 µg GI.1 virus-like particle (VLP) and 150 µg GII.4c VLP, adjuvanted with 500 µg of aluminum hydroxide.
Groups:
- HIL-214: One dose of norovirus GI.1/GII.4c bivalent virus-like particle (VLP) vaccine (HIL-214) (50 µg of GI.1 VLP and 150 µg GII.4c VLP, adjuvanted with 500 µg aluminum hydroxide) by intramuscular injection on Day 1.
Period: Overall Study
Arm/Group | HIL-214
Started | 80
Completed | 77
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, all participants that received trial vaccine (HIL-214).
Arm/Group | HIL-214
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 40
  White | 31
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 80
Weight [Mean (Standard Deviation); unit: kg] | 87.32 (24.573)
Height [Mean (Standard Deviation); unit: cm] | 170.70 (10.822)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.06 (8.358)

OUTCOME MEASURES:

1. Primary Outcome: Primary Immunogenicity for Panel Formation
Description: Serum samples were obtained for validation of the norovirus GI.1 and GII.4c histoblood group antigen (HBGA)-blocking and total immunoglobulin (pan-Ig) assays. The percentage of participants with a predefined seroresponse (≥4-fold rise in antibody concentration from Day 1 to Day 29) to the GI.1 and GII.4c components of HIL-214 and 95% confidence interval are reported.
Time Frame: Day 1 to Day 29
Population: Safety Analysis Set, all participants that received trial vaccine (HIL-214).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HIL-214
Number analyzed (Participants) | 78
Percentage of Participants
  Anti-GI.1 HBGA-blocking seroresponse rate: number analyzed (Participants) | 77
  Anti-GI.1 HBGA-blocking seroresponse rate | 87.0 [77.4 to 93.6]
  Anti-GII.4c HBGA-blocking seroresponse rate: number analyzed (Participants) | 77
  Anti-GII.4c HBGA-blocking seroresponse rate | 72.7 [61.4 to 82.3]
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate: number analyzed (Participants) | 77
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate | 60.5 [48.6 to 71.6]
  Anti-GI.1 pan-Ig seroresponse rate | 98.7 [93.1 to 100]
  Anti-GII.4c pan-Ig seroresponse rate | 91.0 [82.4 to 96.3]
  Anti-GI.1 and GII.4c pan-Ig seroresponse rate | 91.0 [82.4 to 96.3]

2. Secondary Outcome: Adverse Events Leading to Participant Withdrawal From the Trial
Description: Adverse events leading to trial withdrawal were collected throughout the trial.
Time Frame: Day 1 to Day 85
Population: Safety Analysis Set, all participants that received trial vaccine (HIL-214).
Measure: Count of Participants; unit: Participants
Arm/Group | HIL-214
Number analyzed (Participants) | 80
Participants | 0

3. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events Within 7 Days of Vaccine Administration
Description: Assessed solicited local AEs included pain at injection site, redness, swelling, and induration. See AE tables for specifics.
Time Frame: Day 1 to Day 7
Population: Safety Analysis Set, all participants who received trial vaccine (HIL-214).
Measure: Number; unit: percentage of participants
Arm/Group | HIL-214
Number analyzed (Participants) | 79
percentage of participants | 48.1

4. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) Within 7 Days of Vaccine Administration
Description: Assessed solicited systemic AEs included headache, fatigue, myalgia, arthralgia, vomiting, diarrhea, and fever.
Time Frame: Day 1 to Day 7
Population: Safety Analysis Set, all participants who received trial vaccine (HIL-214).
Measure: Number; unit: percentage of participants
Arm/Group | HIL-214
Number analyzed (Participants) | 79
percentage of participants | 55.7

5. Secondary Outcome: Percentage of Participants With at Least One Unsolicited AEs After the Dose of Trial Vaccine
Description: Unsolicited AEs are any local or systemic AEs, as defined by this study, that are not solicited.
Time Frame: Day 1 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | HIL-214
Number analyzed (Participants) | 80
Participants | 7

ADVERSE EVENTS:
Time Frame: Serious adverse events, all-cause mortality and other significant adverse events were assessed for each participant from Day 1 to Day 85
Description: Solicited AE (local and systemic) data was collected for 79 participants.
Arm/Group | HIL-214
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 52/79
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIL-214 (N=79)
Injection site pain (Injury, poisoning and procedural complications) | 35
Redness (Injury, poisoning and procedural complications) | 6
Swelling (Injury, poisoning and procedural complications) | 4
Induration (Injury, poisoning and procedural complications) | 7
Headache (General disorders) | 24
Fatigue (General disorders) | 27
Myalgia (General disorders) | 31
Arthralgia (General disorders) | 11
Vomiting (General disorders) | 4
Diarrhea (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05972733/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT05972733/SAP_001.pdf